CLINICAL TRIAL: NCT02763111
Title: International Multi-center Comparative Randomized Double-blind Placebo-controlled Clinical Trial to Evaluate Efficacy and Safety of Multiple Subcutaneous Injections of BCD-085 in Various Doses in Patients With Active Ankylosing Spondylitis
Brief Title: Clinical Trial to Evaluate Efficacy and Safety of Multiple Subcutaneous Injections of Various Doses of BCD-085 in Patients With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCD-085-3
Record Dates: First submitted 2016-04-03; First posted 2016-05-05 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; interleukin 17; monoclonal antibody
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BCD-085, 40 mg (Experimental): Patient will receive 40 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10, 12.
  Interventions: Drug: BCD-085
- BCD-085, 80 mg (Experimental): Patient will receive 80 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10, 12.
  Interventions: Drug: BCD-085
- BCD-085, 120 mg (Experimental): Patient will receive 120 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10, 12.
  Interventions: Drug: BCD-085
- Placebo (Placebo Comparator): Patient will receive placebo subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10, 12.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BCD-085
  Arms: BCD-085, 120 mg; BCD-085, 40 mg; BCD-085, 80 mg
Other: Placebo
  Arms: Placebo

SUMMARY:
BCD-085-3 is a next step in clinical investigation of BCD-085. BCD-085 is a monoclonal antibody to interleukin 17. During the trial patients with active ankylosing spondylitis will receive 40, 80 or 120 mg of BCD-085 subcutaneously at weeks 0, 1, 2, 4, 6, 8, 10, 12. Efficacy and safety parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age between 18 and 65 years
* Active ankylosing spondylitis according to modified criteria of New York classification (1984), that was diagnosed at least 3 months prior to screening.
* Active disease according to BASDAI (score 4 or more) if nonsteroidal antiinflammatory drugs were used in the last 3 month prior to screening.
* Mean backache intensity equals 4 points or more.
* If patient have had biologic therapy to treat ankylosing spondylitis for at least 3 months, there was no positive results of such treatment or patient revealed intolerance to the drug. This therapy must be discontinued at least 12 weeks before enrollment in the study.
* Female patients have negative urine pregnancy test.
* Patient has no history of tuberculosis.
* Patients have negative results of Diaskintest.
* Patient has no history of alcohol or drug abuse.

Exclusion Criteria:

* Total spinal ankylosis.
* Allergy or intolerance of monoclonal antibodies or any excipients of study drugs.
* Previous receipt of anti-interleukin 17 drugs or anti-interleukin 17 receptor drugs.
* Prior use of two or more biologics to tumor necrosis factor alfa.
* Prior use of two or more biologics to other targets. Previous receipt of monoclonal antibodies if they were cancelled less that in 12 weeks before signing informed consent.
* Patient is taking corticosteroids for up to 4 weeks in a dose more than 10 mg (recalculated to prednisolone) before signing informed consent and during screening, or in a dose less than 10 mg (recalculated to prednisolone) if it was not stable.
* Prior use of disease-modifying antirheumatic drugs including methotrexate, sulfasalazin, chloroquine or hydroxychloroquine for up to 4 weeks before randomization, if their dose was not stable for up to 4 weeks before signing informed consent and during screening.
* Prior use of live or attenuated vaccines for up to 8 weeks before signing informed consent.
* Prior use of alkylating agents for up to 12 months prior to signing informed consent.
* Intraarticular use of corticosteroids for up to 4 weeks before randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Ratio of patients with ASAS20 response after 16 weeks of therapy | Week 16
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 20% or more after 16 weeks of therapy with BCD-085.

SECONDARY OUTCOMES:
Ratio of patients with ASAS20 response after 4, 8, 12 weeks of therapy | Week 4, Week 8, Week 12
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 20% or more after 4, 8, 12 weeks of therapy with BCD-085.
Ratio of patients with ASAS40 response after 4, 8, 12, 16 weeks of therapy | Week 4, Week 8, Week 12, Week 16
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 40% or more after 4, 8, 12, 16 weeks of therapy with BCD-085.
Ratio of patients with ASAS5/6 response after 4, 8, 12, 16 weeks of therapy | Week 4, Week 8, Week 12, Week 16
  Ratio of patients who developed a response in at least 5 of 6 criteria of ankylosing spondylitis assessment score (ASAS) after 4, 8, 12, 16 weeks of therapy with BCD-085.
Mean BASDAI score at screening and after 4, 8, 12, 16 weeks of therapy | Screening, Week 4, Week 8, Week 12, Week 16
  Mean Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score at screening and after 4, 8, 12, 16 weeks of therapy
Mean BASMI score at screening and after 4, 8, 12, 16 weeks of therapy | Screening, Week 4, Week 8, Week 12, Week 16
  Mean Bath Ankylosing Spondylitis Metrology Index (BASMI) score at screening and after 4, 8, 12, 16 weeks of therapy
Mean MASES score at screening and after 4, 8, 12, 16 weeks of therapy | Screening, Week 4, Week 8, Week 12, Week 16
  Mean Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at screening and after 4, 8, 12, 16 weeks of therapy
Mean chest excursion at screening and after 4, 8, 12, 16 weeks of therapy | Screening, Week 4, Week 8, Week 12, Week 16
  Mean chest excursion at screening and after 4, 8, 12, 16 weeks of therapy measured by Cloth Tape Measure Technique
Mean BASFI score at screening and after 4, 8, 12, 16 weeks of therapy | Screening, Week 4, Week 8, Week 12, Week 16
  Mean Bath Ankylosing Spondylitis Functional Index (BASFI) score at screening and after 4, 8, 12, 16 weeks of therapy
Mean ASDAS-CRP score at screening and after 4, 8, 12, 16 weeks of therapy | Screening, Week 4, Week 8, Week 12, Week 16
  Mean Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) score at screening and after 4, 8, 12, 16 weeks of therapy
Mean SF-36 score at screening and after 8 and 16 weeks of therapy | Screening, Week 8, Week 16
  Mean Short Form-36 (SF36) score at screening and after 8, 16 weeks of therapy
Mean pain score during a day at screening and after 1, 2, 4, 8, 12, 16 weeks of therapy | Screening, Week 1, Week 2, Week 4, Week 8, Week 12, Week 16
  Mean pain score during a day at screening and after 1, 2, 4, 8, 12, 16 weeks of therapy measured by Visual Analog Scale for Pain
Proportion of patients with deterioration of roentgenologic signs of sacroileitis after 16 weeks of treatment | Week 16
Mean C-reactive protein concentration at screening and after 4, 8, 12 and 16 weeks of treatment. | Screening, Week 4, Week 8, Week 12, Week 16
Frequency of AE/SAE | 16 weeks
Frequency of local reactions | 16 weeks
Frequency of AE/SAE 3-4 grade CTCAE 4.03 | 16 weeks
Frequency of withdrawals due to AE/SAE | 16 weeks
Cmin | 0 to 168 hours post-dose
  Minimal concentration of BCD-085 in blood after drug injection
AUC (0-168h) | 0 to 168 hours post-dose
  Area under curve from 0 to 168 hours of BCD-085 in blood after drug injection
AUC0-∞ | 0 to 168 hours post-dose
  Area under curve from 0 to infinity of BCD-085 in blood after drug injection
Cmax | 0 to 168 hours post-dose
  Maximal concentration of BCD-085 in blood after drug injection
Тmax | 0 to 168 hours post-dose
  Time before Cmax of BCD-085 is reached in blood after drug injection
Т½ | 0 to 168 hours post-dose
  Half-life of BCD-085 in blood after drug injection
Кel | 0 to 168 hours post-dose
  Elimination rate constant of BCD-085 in blood after drug injection
Cl | 0 to 168 hours post-dose
  Clearance of BCD-085 in blood after drug injection
Proportion of patients who developed binding and neutralizing antibodies to BCD-085 | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JCS BIOCAD

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erdes S, Nasonov E, Kunder E, Pristrom A, Soroka N, Shesternya P, Dubinina T, Smakotina S, Raskina T, Krechikova D, Povarova T, Plaksina T, Gordeev I, Mazurov V, Reshetko O, Zonova E, Eremeeva A, Chernyaeva E, Makulova T, Ivanov R. Primary efficacy of netakimab, a novel interleukin-17 inhibitor, in the treatment of active ankylosing spondylitis in adults. Clin Exp Rheumatol. 2020 Jan-Feb;38(1):27-34. Epub 2019 Apr 16. PMID 31025924